CLINICAL TRIAL: NCT05344807
Title: Role OF Geometric Mean in Estimation OF Differential Renal Function in DMSA Scintigraphy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Shrouk Atef Abdelsalam, resident doctor at Nuclear medicine, Oncology department Sohag university hospital, Sohag University
Other Study IDs: Soh-Med-22-04-06
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Patients Referred for Renal DMSA Scintigraphy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Renal DMSA Scintigraphy — patient injected with Tc99mDMSA then imaged after 2-4 hours by gamma camera

SUMMARY:
Renal scintigraphy is an imaging method that uses small amount of radioactive materials called radiotracers, a Gamma camera and a computer to evaluate kidney functions and its anatomy.

The relative renal function (RRF), expressed as a percent of total renal function, is important in the initial assessment and treatment of patients having renal diseases. RRF has traditionally been measured by radionuclide renal scintigraphies using different tracers for a long time . Different radiopharmaceuticals such as technetium-99m-diethylenetriaminepentaacetic acid (99mTc-DTPA), technetium-99m-dimercaptosuccinic acid (99mTc-DMSA), technetium-99m-mercaptoacetyltriglycine (99mTc-MAG3).

99mTc-DMSA is a static agent that is actively taken up by the proximal and distal renal tubular cells, directly from the peritubular vessels and accumulates in the renal cortex. Its binding level to protein in mammals is 90% which prevents significant glomerular filtration. DMSA renal scan images provide a good definition of the cortical outline, as well as they show the relative distribution of functional tissue.

Determination of the left to right dimercaptosuccinic acid (DMSA) uptake ratio is theoretically one of the easiest quantitative procedures in nuclear medicine. The quantification can be performed on the posterior view, with or without the lateral view for correction of kidney depth. The geometric mean can also be determined using both the anterior and the posterior views.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for renal DMSA scintigraphy
* Patients aging 2 to 70 years

Exclusion Criteria:

* Single kidney patients
* Patients with a major uncontrollable medical illness.

Ages: 2 Years to 70 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: • Patients referred for renal DMSA scintigraphy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
geometric mean of both anterior and posterior views of gamma camera | 6 months
  . We evaluate the discrepancy between function measured by conjugate anterior and posterior views in relationship to posterior view in DMSA scan .

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arteaga MV, Caballero VM, Rengifo KM. Dosimetry of 99mTc (DTPA, DMSA and MAG3) used in renal function studies of newborns and children. Appl Radiat Isot. 2018 Aug;138:25-28. doi: 10.1016/j.apradiso.2017.07.054. Epub 2017 Jul 28. PMID 28781122
- [Background] Hervas I, Marti JF, Gonzalez A, Ruiz JC, Alonso J, Bello P, Manzano F, Torres I, Mateo A. Is the depth correction using the geometric mean really necessary in a 99Tcm-DMSA scan in the paediatric population? Nucl Med Commun. 2001 May;22(5):547-52. doi: 10.1097/00006231-200105000-00013. PMID 11388577
- [Background] Miyazaki C, Harada H, Shuke N, Okizaki A, Miura M, Hirano T. (99m)Tc-DTPA dynamic SPECT and CT volumetry for measuring split renal function in live kidney donors. Ann Nucl Med. 2010 Apr;24(3):189-95. doi: 10.1007/s12149-010-0349-y. Epub 2010 Mar 9. PMID 20213340